CLINICAL TRIAL: NCT04669158
Title: A Pilot Study to Treat Adults With Non-Alcoholic Steatohepatitis With Oral Idebenone
Brief Title: Study of Oral Idebenone to Treat Non-Alcoholic Steatohepatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Natalie Torok, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 52212; R21DK111217 (NIH)
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Non Alcoholic Steatohepatitis; Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Idebenone (Experimental): Participants will take Idebenone 200 mg for 48 weeks, with study visits in clinic for physical and laboratory assessments at weeks 0, 2, 4, 12, 24, 36, and 48 weeks during treatment period and at 4, and 12 weeks after the last dose.
  Interventions: Drug: Idebenone
- Placebo (Placebo Comparator): Participants will take Placebo for 48 weeks, with study visits in clinic for physical and laboratory assessments at weeks 0, 2, 4, 12, 24, 36, and 48 weeks during treatment period and at 4, and 12 weeks after the last dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Idebenone — Idebenone, initially 200mg by mouth (P.O.) once a day for 2 weeks, then 200 mg twice a day for 2 weeks, then 200 mg three times per day for the remainder of the study will be used.
  Arms: Idebenone
Drug: Placebo — Placebo to match Idebenone once a day for 2 weeks, then twice a day for 2 weeks, then three times per day for the remainder of the study will be used.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled phase 1/2a study to investigate the safety and tolerability of Idebenone in patients 18 years of age or older with non-alcoholic steatohepatitis, with stage 1-3 fibrosis. As secondary end point target engagement and fibrosis improvement will be assessed.

DETAILED DESCRIPTION:
This is a prospective phase 1/2a, randomized, double-blinded, placebo-controlled, single center study of safety and efficacy of oral idebenone in adults 18 years of age or older with non-alcoholic steatohepatitis (NASH). Following IRB approval and written informed consent, 45 participants will be enrolled in the study and randomized in a 1:2 ratio on REDCap data capturing software. Participants will be randomized to two groups and receive the following tablets: placebo, idebenone at escalating doses of 200mg by mouth (P.O.) once a day for 2 weeks, then 200 mg twice a day for 2 weeks, then 3 times per day for the remainder of the study (up to 48 weeks). Monitoring and safety evaluation will continue for 12 weeks after the final dose. The study will investigate the safety and tolerability as primary end point and assess target engagement and fibrosis improvement as secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* 1) Male or non-pregnant/ non-lactating women ≥ 18 years of age
* 2) Diagnosis of NASH: NAFLD activity score (NAS) of 4 or greater with a score of 1 for each of the following (steatosis scored 0-3, lobular inflammation scored 0-3, ballooning scored 0-2):

  * Steatosis
  * Lobular inflammation
  * Hepatocyte ballooning 3) Fibrosis (Ishak fibrosis score ≥1 on liver biopsy) within 6 months of enrollment with MELD<10, or based on MRE

Exclusion Criteria:

* Presence of any other form of liver disease, including viral hepatitis, autoimmune hepatitis, alcoholic liver disease, genetic causes of chronic liver disease):
* Subjects with other etiologies of chronic liver disease, such as chronic hepatitis B and C; autoimmune hepatitis; and inherited liver disease.
* ALT>300 U/l
* Total serum bilirubin ≥ to 1.3 mg/dL (Gilbert's Syndrome patients excepted)
* International Normalized Ratio (INR) ≥ 1.3
* MELD>10
* Serum creatinine >2.0mg/dl
* Known alcohol abuse or alcohol use disorder:

  * >20 g/day for women
  * >30 g/day for men
* Active substance abuse
* Any medical condition that prevents MRE, MR-PDFF
* Platelet count ≤100//mm3
* Decompensated cirrhosis
* Hemoglobin <11 g/dl in females or <12 g/dl in males
* Presence/history of HCC
* History of liver transplantation
* History of bariatric surgery
* History of inflammatory bowel disease
* History of cardiovascular disease, long QT syndrome.
* Subjects who have participated in investigational drug trials and took any investigational drugs within 60 days prior to the first dose of Idebenone. History of receiving other investigations drug within 30 days prior to enrollment
* Any concerns regarding compliance by enrolling physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Week 60: Assessment of AEs
  Number of Participants with Treatment-Related Adverse Events (Assessed by CTCAE v4.0, including abnormal Physical exams and abnormal laboratory tests results will be reported.

SECONDARY OUTCOMES:
Change in fibrosis stage | Week 48: fibrosis change
  Number of Participants with change in fibrosis stage

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Torok, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Digestive Health Center, Stanford University, Redwood City, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No